CLINICAL TRIAL: NCT04868123
Title: Pilot Study of Mindfulness Meditation and Transcutaneous Nerve Stimulation (TENS) in Persons Living With HIV-related Peripheral Neuropathy
Brief Title: Effects of TENS and Mindfulness Meditation in Persons With HIV-related Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, David Kietrys, Associate Professor, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2020003234
Record Dates: First submitted 2021-04-25; First posted 2021-04-30 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: peripheral neuropathy; pain; TENS; Mindfulness Meditation
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Pain | interventions — Transcutaneous Electric Nerve Stimulation; Mindfulness

STUDY DESIGN:
Intervention Model Description: randomized controlled interventional pilot with 3 groups (2 treatment groups and 1 control group)
Who Masked: Outcomes Assessor
Masking Description: co-investigators involved with measurement for the interventional phase will not know which of the 3 groups a participant was randomized to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Mindfulness Meditation (Experimental): 6 weeks of daily mindfulness meditation (guided by audio recordings) performed at home
  Interventions: Behavioral: Mindfulness Meditation
- Transcutaneous nerve stimulation (TENS) (Experimental): 6 weeks of daily TENS treatment performed at home
  Interventions: Device: Transcutaneous Nerve Stimulation (TENS)
- Usual Care (No Intervention): Usual care (no additional treatment)

INTERVENTIONS:
Device: Transcutaneous Nerve Stimulation (TENS) — Transcutaneous nerve stimulation (TENS) is a simple home base treatment to manage pain. It involves electrical current applied to the skin through self-adhering electrodes, using a TENS3000 device (TENSPros.com).
  Arms: Transcutaneous nerve stimulation (TENS)
Behavioral: Mindfulness Meditation — Mindfulness mediation is a guided mediation process to improve awareness of being present in the moment.
  Arms: Mindfulness Meditation

SUMMARY:
This study is to explore the effects of transcutaneous nerve stimulation (TENS) and mindfulness meditation in persons living with HIV (PLHIV) and painful neuropathy in the feet.

DETAILED DESCRIPTION:
The overall goal of this study is to conduct an interventional pilot trial of mindfulness meditation and transcutaneous nerve stimulation (TENS) to mitigate the symptoms and improved function in persons living with HIV (PLHIV) and painful neuropathy in the feet. .

The investigators aim to determine the feasibility and effects of (1) mindfulness meditation or (2) transcutaneous nerve stimulation (TENS) on clinical and functional outcomes in participants with HIV-associated painful distal sensory polyneuropathy in the feet. This aim will be achieved with a randomized control pilot trial with 3 groups: TENS group, Mindfulness Mediation Group, and Usual Treatment (Control) group. The interventions will be performed at home over a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HIV infection currently treated with antiretroviral therapy (ART)
* cluster of differentiation 4 cell (CD4 cell) count of at least 200 cells/mm3
* 18-64 years of age
* able to read and write in English
* means to travel to a study site
* presence of peripheral neuropathy symptoms in feet
* average daily self-reported pain in the feet of at least 3/10 on a 0-10 numerical pain scale
* pain in the feet present for at least the past 3 months
* no changes in medications used to manage pain in the past 4 weeks
* no use of TENS or mindfulness meditation in the prior 6 months
* availability of a mobile phone to receive text messages over the course of the intervention period

Exclusion Criteria:

* current opportunistic infection(s)
* cluster of differentiation 4 cell (CD4 cell) count <200 cells/mm3
* dementia
* uncontrolled psychiatric disorder
* wounds or sores on the feet
* musculoskeletal or neurological conditions (other than distal sensory neuropathy) that may affect gait
* pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain Intensity at 7 weeks | Week 0 and Week 7
  Responses to questions on the Brief Pain Inventory Pain Intensity subscale used to generate pain intensity score. Minimum score=0; maximum score=10; higher score=worse outcome.
Change from Baseline Pain Interference at 7 weeks | Week 0 and Week 7
  Responses to questions on the Brief Pain Inventory Pain Interference subscale used to generate pain interference score. Minimum score=0; maximum score=10; higher score=worse outcome.

SECONDARY OUTCOMES:
Change from Baseline Pain Pressure Threshold at 7 weeks | Week 0 and Week 7
  Pain pressure threshold (expressed in pounds or kilograms of force) at lower extremity landmarks via use of a digital algometer.
Change from Baseline Gait Characteristics at 7 weeks | Week 0 and Week 7
  Temporal and spatial characteristics of gait (walking velocity, step length, step time, stride width, cadence, foot-fall area) as captured with a ZENO instrumented walkway
Change from Baseline Walking Endurance at 7 weeks | Week 0 and Week 7
  Walking endurance as measured with the 6-Minute Walk test (distance walked over span of 6 minutes).
Change in Baseline Physical Performance at 7 weeks | Week 0 and Week 7
  Physical performance score generated via the Short Physical Performance Battery. (SPPB). SPPB procedures generate a total score reflective of physical performance. Minimum score=0; maximum score=12; lower score=worse outcome.
Change from Baseline Whole Body Strength at 7 weeks | Week 0 and Week 7
  Mid-thigh pull test will be used to generate a score expressed as force in pounds or kilograms that is reflective of whole body strength.
Change from Baseline Physical Activity at 7 weeks | Week 0 and Week 7
  Physical activity characteristics: (1) over a span of 5 days captured via a wrist-band style Actigraph activity monitor, and (2) self-reported physical activity over past 7 days using the International Physical Activity Questionnaire - Short Form
Change from Baseline Mental Quality of Life (QOL) at 7 weeks | Week 0 and Week 7
  Mental Health Summary Score generated via responses on the Medical Outcomes Study HIV Health Survey (MOS-HIV). Minimum score=0; maximum score=100; lower score=worse outcome.
Change from Baseline Physical Quality of Life (QOL) at 7 weeks | Week 0 and Week 7
  Physical Health Summary Score generated via responses on the Medical Outcomes Study HIV Health Survey (MOS-HIV). Minimum score=0; maximum score=100; lower score=worse outcome.
Change from Baseline Depression at 7 weeks | Week 0 and Week 7
  Self-reported depression as determined by the depression subscale of the Hospital Depression and Anxiety Scale. Minimum score=0; maximum score=21; higher score=worse outcome.
Change from Baseline Anxiety at 7 weeks | Week 0 and Week 7
  Self-reported anxiety as determined by the anxiety subscale of the Hospital Depression and Anxiety Scale. Minimum score=0; maximum score=21; higher score=worse outcome.
Change from Baseline Catastrophizing Behaviors at 7 weeks | Week 0 and Week 7
  Self-reported catastrophizing behaviors using with the Pain Catastrophizing Scale. Minimum score=0; maximum score=52; higher score=worse outcome.
Change from Baseline Resilience behaviors at 7 weeks | Week 0 and Week 7
  Self-reported resilience using the 6-item Brief Resilience Scale. Minimum score=1; maximum score=5; lower score=worse outcome.
Change from Baseline Pain Medication Use at 7 weeks | Week 0 and Week 7
  Self-report of use of pain medication base on responses to a study-specific questionnaire
Satisfaction with Study Experiences | week 7
  Self-reported satisfaction with the study parameters and study experiences using a study-specific questionnaire
Adherence to Home-based Treatment (TENS and Mindfulness Meditation groups) | week 6
  Tracking of adherence to home based intervention (number of sessions per week completed and total number of sessions completed over 6 weeks) via direct communication with participants

CONTACTS AND LOCATIONS:
Overall Officials: David M Kietrys, PhD, Principal Investigator — Rutgers
Locations (2):
- United States (2):
  - Rutgers Physical Therapy Program, Blackwood, New Jersey
  - Rutgers Physical Therapy Program, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04868123/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT04868123/ICF_001.pdf